CLINICAL TRIAL: NCT03947242
Title: Neoadjuvant Study of Pyrotinib in Combination With Trastuzumab Plus Vinorelbine in Trastuzumab-refractory HER2-Positive Early Stage or Locally Advanced Breast Cancer Patients.
Brief Title: Neoadjuvant Study of Pyrotinib and Trastuzumab Plus Vinorelbine in Trastuzumab-refractory HER2-Positive Breast Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-NeoBC-HN003
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: HER2 Positive Breast Cancer
Keywords: Trastuzumab-refractory
MeSH Terms: interventions — pyrotinib; Trastuzumab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib + trastuzumab +Vinorelbine (Experimental): Pyrotinib in Combination With Trastuzumab Plus Vinorelbine
  Interventions: Drug: Pyrotinib and Trastuzumab plus Vinorelbine

INTERVENTIONS:
Drug: Pyrotinib and Trastuzumab plus Vinorelbine — Pyrotinib:400mg orally daily Trastuzumab:8mg/kg ivgtt load followed by 6mg/kg ivgtt 3-weekly for a total of 4 cycles Vinorelbine :25mg/m2 ivgtt 3-weekly for a total of 4 cycles,d1 d8

SUMMARY:
This study is a single-arm, prospective, open label clinical study for evaluating the efficacy and safety of neoadjuvant pyrotinib and trastuzumab plus Vinorelbine given as neoadjuvant treatment in Trastuzumab-refractory HER2 positive early stage or locally advanced breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant therapy is the standard treatment for locally advanced breast cancer and is used to reduce tumors to make them operable, and to increase breast-conserving rates. In recent years, the anti-HER2 treatment mode, which is double-blocked by a combination of dual-targeted drugs, has obtained clinical approval in adjuvant therapy and neoadjuvant therapy. Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. Based on previous clinical studies, we designed the study to explore the possibility of Pyrotinib in combination with Trastuzumab plus Vinorelbine given as neoadjuvant treatment in HER2 positive early stage or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. female patients, 18 years ≤ age ≤ 75 years. 2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1. 3. Histologically confirmed invasive breast cancer:early stage or locally advanced,Primary tumour greater than 2 cm diameter 4. HER2 positive (HER2+++ by IHC or FISH+) 5. Subjects received neoadjuvant therapy with trastuzumab 2 weeks post-imaging evaluation Patients with a price of PD or SD. 6. Known hormone receptor status. 7. Required laboratory values including following parameters: ANC: ≥ 1.5 x 10^9/L;Platelet count: ≥ 100 x 10^9/L;Hemoglobin: ≥ 9.0 g/dL;Total bilirubin: ≤ 1.5 x upper limit of normal (ULN);ALT and AST: ≤ 1.5 x ULN (or ≤ 5×ULN in patients with liver metastases);BUN and creatine clearance rate: ≥ 50 mL/min;LVEF: ≥ 50%;QTcF: < 470 ms for female and < 450 ms for male. 8. Signed the informed consent form prior to patient entry.

Exclusion Criteria:

- 1. metastatic disease (Stage IV) or inflammatory breast cancer. 2. Previous or current history of malignant neoplasms, except for curatively treated:Basal and squamous cell carcinoma of the skin,Carcinoma in situ of the cervix.

3. clinically relevant cardiovascular disease:Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110); 4. Unable or unwilling to swallow tablets.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | [Time Frame: Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months
  Objective Response Rate

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | Time Frame: through study completion, an average of 1 year
  Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery evaluated
EFS | Time Frame: Following surgery until Year 5
  Event-free survival
DFS | Time Frame: Following surgery until Year 5
  Disease-free Survival
DDFS | Time Frame: Following surgery until Year 5
  Distance Disease-free Survival

CONTACTS AND LOCATIONS:
Overall Officials: xiuchun Chen, Principal Investigator — Study Principal Investigator Henan Cancer Hospital